CLINICAL TRIAL: NCT01532492
Title: Validation of the Western Ontario Rotator Cuff Index in Patients With Arthroscopic Rotator Cuff Repair
Acronym: WORC
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Ronald Wessel, Principal investigator, St. Antonius Hospital
Other Study IDs: LTME/Z-11.19/WORC
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Rotator Cuff Lesion; Disorder of Rotator Cuff; Other Instability, Shoulder
Keywords: Questionnaire; WORC; Rotator cuff; Reliability; Validity; Responsiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Rotator cuff repair group: Patients undergoing an arthroscopic rotator cuff repair
- DRC without rupture: Disorders of the rotator cuff without rupture
- Shoulder instability: Shoulder instability

SUMMARY:
Arthroscopic rotator cuff repair is described as being a successful procedure. These results are often derived from clinical general shoulder examinations, which are then classified as 'excellent', 'good', 'fair' or 'poor'. However, the cut-off points for these classifications vary and sometimes modified scores are used.

Arthroscopic rotator cuff repair is performed to improve quality of life. Therefore, disease specific health-related quality of life patient-administered questionnaires are needed. The WORC is a quality of life questionnaire designed for patients with disorders of the rotator cuff. The score is validated for rotator cuff disease, but not for rotator cuff repair specifically.

The aim of this study is to investigate reliability, validity and responsiveness of WORC in patients undergoing arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
An approved translation of the WORC into Dutch is used. In this prospective study three groups of patients are used: 1.Arthroscopic rotator cuff repair; 2.Disorders of the rotator cuff without rupture; 3.Shoulder instability.

The WORC, SF-36 and the Constant Score are obtained twice before therapy is started to measure reliability and validity. Responsiveness is tested by obtaining the same tests after therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* written informed consent
* diagnosis for group 1, 2 or 3

Exclusion Criteria:

* lack of understanding the Dutch language
* not able to complete questionnaires independently
* additional shoulder pathology like adhesive capsulitis, AC-pathology and osteoarthritis
* previous shoulder surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients undergoing arthroscopic rotator cuff repair. These patients have a clinical suspicion of a symptomatic rotator cuff tear and a partial or full thickness lesion seen on MRI or Ultrasound and confirmed during the arthroscopic repair procedure.
  2. Patients diagnosed as having non-Ruptured DRC. They have a clinical suspicion of DRC and no rupture of the rotator cuff on MRI or Ultrasound.
  3. Patients will be diagnosed with shoulder instability
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Reliability of the WORC | 6 months
  Reliability of the WORC is tested by comparing the results at T0 with T1. T1 is planned 2-3 weeks after T0, because we expect that the symptoms do not change between these two moments and the time span is large enough to forget initial responses to the questions. In order to signal change in severity of the symptoms, at both moments patients are asked to rate their shoulder hindrance. To determine test-retest reliability, intraclass correlation coefficients (ICC) are used.

SECONDARY OUTCOMES:
Criterion validity of the WORC | 6 months
  Criterion validity is measured by comparing WORC with a general quality of life questionnaire (SF-36) and a commonly used clinical shoulder score (Constant Score) both at T0 and T1. Bland Altman plots will be used to estimate 95% boundaries of concurrence.
Responsiveness of the WORC | 6 months
  Responsiveness will be determined by calculating the standardized response means and effect sizes on T0 and T2 scores on WORC, SF-36 and Constant scores for the subgroups.
Differentiation between patient groups | 6 months
  A comparison of WORC scores between the three distinct groups is made, to see whether WORC scores can differentiate between them. WORC scores will be compared with SF-36 to investigate whether the noted differences correlate with notable clinical differences and can be expressed as MCID's (minimal clinical important differences).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald N Wessel, MD, Principal Investigator — St. Antonius Hospital; Henk van Mameren, PhD, MD, Principal Investigator — Department of Epidemiology, Caphri research school, Maastricht University; Rob A de Bie, PhD, MA, RPt, Principal Investigator — Department of Epidemiology, Caphri research school, Maastricht University
Locations (1):
- Department of Orthopedics, St. Antonius Hospital, Nieuwegein, Netherlands

REFERENCES:
- [Derived] Wessel RN, Wolterbeek N, Fermont AJ, van Mameren H, Sonneveld H, Griffin S, de Bie RA. The conceptually equivalent Dutch version of the Western Ontario Rotator Cuff Index (WORC)(c). BMC Musculoskelet Disord. 2013 Dec 21;14:362. doi: 10.1186/1471-2474-14-362. PMID 24359231